CLINICAL TRIAL: NCT02740842
Title: A Follow-up Study on the Sustained Impact of Alive & Thrive Behavior Change Communication Interventions on Infant and Young Child Feeding Practices in Bangladesh
Brief Title: A Follow-up Study on the Sustained Impact of Alive & Thrive Interventions on Infant and Young Child Feeding Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IFPRI_1
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2017-02

CONDITIONS: Breastfeeding; Complementary Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-intensive group (Active Comparator): Essential Health Care (EHC) only This arm is the basic comparison arm, which will receive the standard package of health services offered through BRAC's essential health care (basic antenatal care, basic counseling on health and nutrition through health worker home visits. In addition, a nationwide mass media campaign on IYCF practices will ensure exposure to some messages about IYCF behaviors in this arm.
  Interventions: Behavioral: Mass media
- Intensive group (Experimental): Interpersonal behavioral change communication This arm will have a behavior change communications intervention to improve infant and young child feeding practices. The intervention will be delivered primarily by the frontline health workers who will visit mothers in their homes and counsel them on essential IYCF practices.
  In addition, a nationwide mass media campaign on IYCF practices will ensure exposure to some messages about IYCF behaviors in this arm.
  Interventions: Behavioral: Interpersonal behavioral change communication; Behavioral: Mass media

INTERVENTIONS:
Behavioral: Interpersonal behavioral change communication — This arm includes home visits to mothers with infants and young children. Frontline health workers will counsel and support mothers in relation to breastfeeding and complementary feeding practices
  Arms: Intensive group
Behavioral: Mass media — A nationwide mass media campaign of TV and radio spots on infant and young child feeding practices will be aired in 2011, 2012 and 2013. All intervention arms will be exposed to this campaign.

SUMMARY:
Alive & Thrive (A&T) is a multi-year initiative to improve infant and young child feeding (IYCF) practices. During Phase 1 (A&T-1, 2009-2014), funded by the Bill & Melinda Gates Foundation, A&T aimed to reduce undernutrition and death caused by suboptimal IYCF practices in three countries - Bangladesh, Ethiopia, and Viet Nam.

In 2014, IFPRI in collaboration with DATA conducted the endline survey in Bangladesh. The overall findings of the evaluation indicate that A&T's work in Bangladesh is a remarkable success story of scaling up what has been challenging to date in the field of nutrition: complex, high intensity and at-scale behavior change communications interventions.

In 2016, a follow up study will be conducted to determine the sustained impacts on IYCF practices, expansion of operations and promoted practices into new areas, and diffusion of IYCF information, two years after the termination of external project support.

DETAILED DESCRIPTION:
Alive & Thrive (A&T) is a multi-year initiative to improve infant and young child feeding (IYCF) practices. During Phase 1 (A&T-1, 2009-2014), funded by the Bill & Melinda Gates Foundation, A&T aimed to reduce undernutrition and death caused by suboptimal IYCF practices in three countries - Bangladesh, Ethiopia, and Viet Nam.

A&T-1 strategies in Bangladesh were designed to support improvements in IYCF in three key ways: 1) improving policy and regulatory environments (advocacy); 2) shaping IYCF demand and practice (community-based interventions); and 3) increasing supply, demand, and use of high quality complementary foods (private sector engagement). In addition, a communications component was integrated into each of these focus areas to support their activities.

In 2014, IFPRI in collaboration with DATA conducted the endline survey. The overall findings of the evaluation indicate that A&T's work in Bangladesh is a remarkable success story of scaling up what has been challenging to date in the field of nutrition: complex, high intensity and at-scale behavior change communications interventions. This is demonstrated by a series of findings on reach of the interpersonal counseling interventions and the mass media, as well as attributable improvements in several critical indicators. During the intervention period, A&T facilitated the training of over 75,000 frontline workers and health providers across the country. The program model reached large scale with an estimated 1.7 million mothers of children under 2 years in 50 sub-districts. The mass media intervention operated at a national level and through national television channels. Compared to the 2010 baseline survey, improvements were seen in several key IYCF practices that are attributable to A&T intensive package of interventions. Specifically, large significant impacts were seen on two key breastfeeding indicators: EBF (DID impact estimates: 36.9 percentage point-pp) and early initiation of BF (DID 19.4 pp). Similarly, large significant impact were seen in minimum dietary diversity (DID 16.3 pp), minimum meal frequency (DID 14.7 pp), minimum acceptable diet (DID 22.0 pp), and consumption of iron rich food (DID 24.6 pp).

In 2016, a follow up study will be conducted to determine the sustained impacts on IYCF practices, expansion of operations and promoted practices into new areas, and diffusion of IYCF information, two years after the termination of external project support. Because achievements related to service delivery and outcomes are intended to be sustained in the intervention areas and even expanded to other areas where BRAC's Essential Health Care program operates, including the comparison areas, this study aims to examine elements in both the original intervention and comparison areas.

This study focuses on the follow-up survey of the BRAC community-based model. The study research questions include:

Sustained impacts

1. To what extent are IYCF knowledge and practices sustained in the intervention areas?
2. To what extent is exposure to IYCF and nutrition behavior change communications sustained in the intervention areas?

Expanded operations and reach 1) To what extent has exposure to IYCF and nutrition behavior change communications been expanded (i.e. in comparison areas)?

Diffusion of information

1) To what extent is IYCF information diffused through social networks or by other sources (i.e. other than BRAC frontline workers)?

ELIGIBILITY:
Inclusion Criteria:

* Women with children <24 months of age

Exclusion Criteria:

* Age <18
* Mental disorders that cannot understand and answer the questions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2400 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding (EBF) among children 0-6 months of age | 2 years after endline
  The proportion of infants less than 6 months who have been exclusively breastfed on the day preceding the interview
Early initiation of breastfeeding | 2 years after endline
  The proportion of newborns aged less than 24 months who were breastfed within 1 hour of birth.
Complementary feeding among children 6-23.9 months of age | 2 years after endline
  Complementary feeding indicators that include timely introduction of complementary foods (infants 6-8 months), dietary diversity (consumed at least 4 food groups), minimum meal frequency, will be measured using questionnaire.

SECONDARY OUTCOMES:
Extension of exposure to IYCF and nutrition behavioral change communication | 2 years after endline
  Proportion of mothers with children <2 years exposed to IYCF and nutrition messages
Diffusion of IYCF information though social network | 2 years after endline
  Number of sources that provide IYCF information or messages
Knowledge of infant and young child feeding | 2 years after endline
  Proportion of mothers report correct knowledge on breastfeeding and complementary feeding based on questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- International Food Policy Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nguyen PH, Frongillo EA, Kim SS, Zongrone AA, Jilani A, Tran LM, Sanghvi T, Menon P. Information Diffusion and Social Norms Are Associated with Infant and Young Child Feeding Practices in Bangladesh. J Nutr. 2019 Nov 1;149(11):2034-2045. doi: 10.1093/jn/nxz167. PMID 31396621
- [Derived] Kim SS, Nguyen PH, Tran LM, Sanghvi T, Mahmud Z, Haque MR, Afsana K, Frongillo EA, Ruel MT, Menon P. Large-Scale Social and Behavior Change Communication Interventions Have Sustained Impacts on Infant and Young Child Feeding Knowledge and Practices: Results of a 2-Year Follow-Up Study in Bangladesh. J Nutr. 2018 Oct 1;148(10):1605-1614. doi: 10.1093/jn/nxy147. PMID 30169665